CLINICAL TRIAL: NCT01786824
Title: Preventing Nephropathy Induced by Iodinated Contrast Media in Patients With Renal Impairment: a Randomized Trial Evaluating the Effectiveness of Two Hydration Strategies and L-carnitine Administration
Brief Title: Preventing Contrast-induced Nephropathy: Evaluating Hydration Strategies and L-carnitine Administration
Acronym: CinBiCarn
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Patient pathway has become infeasible due to pressure for shorter hospital stays. Not enough inclusions.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2012/PR-03; 2012-004134-42 (EudraCT Number)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Acute Kidney Injury; Renal Insufficiency
Keywords: contrast induced nephropathy; hydration strategy; L-carnitine
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bicarbonate (Experimental): The patients included in this arm will be administered a hydration regime for the prevention of contrast-induced nephropathy containing sodium bicarbonate.
  Intervention: Hydration strategy using sodium bicarbonate Intervention: Coronarography
  Interventions: Drug: Hydration strategy using sodium bicarbonate; Procedure: Coronarography
- Saline (Active Comparator): The patients included in this arm will be administered a hydration regime for the prevention of contrast-induced nephropathy using sodium chloride solution.
  Intervention: Hydration strategy using saline Intervention: Coronarography
  Interventions: Drug: Hydration strategy using saline; Procedure: Coronarography
- Bicar + L-Carnitine (Experimental): The patients included in this arm will be administered a hydration regime for the prevention of contrast-induced nephropathy containing sodium bicarbonate. They will also receive an oral L-carnitine solution on days -1, 0, 1 to 7.
  Intervention: Hydration strategy using sodium bicarbonate Intervention: L-carnitine Intervention: Coronarography
  Interventions: Drug: Hydration strategy using sodium bicarbonate; Drug: L-carnitine; Procedure: Coronarography
- Saline + L-carnitine (Experimental): The patients included in this arm will be administered a hydration regime for the prevention of contrast-induced nephropathy using sodium chloride solution. They will also receive an oral L-carnitine solution on days -1, 0, 1 to 7.
  Intervention: Hydration strategy using saline Intervention: L-carnitine Intervention: Coronarography
  Interventions: Drug: Hydration strategy using saline; Drug: L-carnitine; Procedure: Coronarography

INTERVENTIONS:
Drug: Hydration strategy using saline — For 12 hours preceding the coronarography, and for 12 following the coronarography, 0.9% sodium chloride at 1 ml/kg/h is administered via a slow intravenous perfusion.
  Other Names: Sodium chloride hydration
  Arms: Saline; Saline + L-carnitine
Drug: Hydration strategy using sodium bicarbonate — For 4-6 hours before the coronarography and for 4-6 hours after the coronarography, 500 ml of isotonic sodium bicarbonate solution (1.4%) will be administered via a slow intravenous solution.
  Arms: Bicar + L-Carnitine; Bicarbonate
Drug: L-carnitine — Before the coronarography (D-1), 1 gram of L-carnitine is administered via an oral solution that can be diluted in a small amount of sugar water if necessary. This administration corresponds to the beginning of a hydration protocol.
  For days 0 to 7 after the coronarography, patients are administered an oral L-carnitine solution (3 grams of L-carnitine per day). The latter may be diluted in a small amount of sugar water if needed.
  Arms: Bicar + L-Carnitine; Saline + L-carnitine
Procedure: Coronarography — All patients included in this study are programmed for a coronarography with injection of contrast material (either iodixanol or ioxaglate). The day of coronarography = Day 0.

SUMMARY:
The general objective of this open, pilot study is to characterize biological parameters related to acute kidney injury among patients undergoing a programmed coronarography with injection of contrast material. The study focuses on two main factors that may influence acute kidney injury: (1) sodium chloride hydration strategy versus sodium bicarbonate hydration strategy and (2) presence of oral L-carnitine treatment versus absence of oral L-carnitine treatment. We will also test for a potential interaction between these two factors.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is scheduled for a coronarography
* The patient can come back to the hospital on days 2 and 7 after the coronarography for follow up
* The patient has moderate to severe renal insufficiency (glomerular filtration rate < 60 ml / min / 1.73 m^2)
* The patient has not had any oral antidiabetic treatments, or diuretic treatments, within 48 hours preceding the coronarography
* Lack of treatment with ACE inhibitors or ARA2 24 hours prior to coronary

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by another study
* The patient is under judicial protection
* The patient is under any kind of guardianship
* The patient refuses to sign the consent form
* It is impossible to correctly inform the patient
* The patient is unable to participate in follow-up visits at days 2 and 7 after the coronarography
* The patient is pregnant or breastfeeding
* The patient is taking L-carnitine
* The patient has a contra indication for a treatment used in this study
* Acute heart failure
* Infarction, acute phase
* Hemodialysis patient
* Myeloma
* Epileptic patient treated with Depakine (valproic acid) (carnitine can lower epilepsy-related thresholds by speeding up the metabolism of Depakine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in glomerular filtration rate | baseline versus 48 hours after contrast injection
  The change in MDRD glomerular filtration rate before coronarography, and 48 hours after the injection of contrast material.

SECONDARY OUTCOMES:
Contrast induced nephropathy? | Day 2
  The presence/absence of contrast induced nephropathy, defined by the presence of at least one of the following:
  1. a >= 25% increase in creatinemia as compared to baseline
  2. an absolute increase >= 44 µmol/L in creatinemia as compared to baseline
  3. a decrease >= 25% in glomerular filtration rate as compared to baseline
Contrast induced nephropathy? | Day 3
  The presence/absence of contrast induced nephropathy, defined by the presence of at least one of the following:
  1. a >= 25% increase in creatinemia as compared to baseline
  2. an absolute increase >= 44 µmol/L in creatinemia as compared to baseline
  3. a decrease >= 25% in glomerular filtration rate as compared to baseline
Contrast induced nephropathy? | Day 7
  The presence/absence of contrast induced nephropathy, defined by the presence of at least one of the following:
  1. a >= 25% increase in creatinemia as compared to baseline
  2. an absolute increase >= 44 µmol/L in creatinemia as compared to baseline
  3. a decrease >= 25% in glomerular filtration rate as compared to baseline
Change in creatinemia | baseline versus Day 2
  The brute change in creatinemia between baseline and Day 2
Change in creatinemia | baseline versus Day 3
  The brute change in creatinemia between baseline and Day 3
Change in creatinemia | baseline versus Day 7
  The brute change in creatinemia between baseline and Day 7
% Change in creatinemia | baseline versus Day 2
  % change in creatinemia between baseline and Day 2
% Change in creatinemia | baseline versus Day 3
  % change in creatinemia between baseline and Day 3
% Change in creatinemia | baseline versus Day 7
  % change in creatinemia between baseline and Day 7
Change in glomerular filtration rate compared to baseline | baseline versus Day 2
  Change in glomerular filtration (MDRD; ml/min/1.73m^2) rate compared to baseline
Change in glomerular filtration rate compared to baseline | baseline versus Day 3
  Change in glomerular filtration (MDRD; ml/min/1.73m^2) rate compared to baseline
Change in glomerular filtration rate compared to baseline | baseline versus Day 7
  Change in glomerular filtration (MDRD; ml/min/1.73m^2) rate compared to baseline
Quantity of contrast material injected / glomerular filtration rate | Day 0 - just after coronarography
Quantity of iodine injected / glomerular filtration rate | Day 0, just after coronarography
Hemodialysis necessary? | Day 7
  Was hemodialysis required for the patient? yes/no
Mortality | Day 7
  The patient passed away during the study. yes/no
Change in serum ngal | baseline (just before coronarography) versus 4 hours after contrast injection
  The change in serum ngal (neutrophil gelatinase associated lipocalin) between baseline and 4 hours after the injection of contrast material.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Reboul, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (5):
- France (5):
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard
  - CHU d'Angers - Hôtel-Dieu, Angers
  - CH d'Avignon - Centre Hospitalier Henri Duffaut, Avignon
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CH de Perpignan - Hôpital Saint Jean, Perpignan